CLINICAL TRIAL: NCT05895253
Title: Safety and Efficacy of Vibro-tactile Feedback for Patients Who Underwent Lower Limb Amputation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment rate of patients was not sufficient during COVID-19; problems with the quality of the primary outcome data collected
Sponsor: Ludwig Boltzmann Institute for Traumatology - The research center in cooperation with AUVA (Other Government)
Collaborators: Saphenus Medical Technology GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: IPS002
Record Dates: First submitted 2023-05-19; First posted 2023-06-08 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Amputation of Lower Limb Below Knee; Unilateral
Keywords: lower limb amputation; somatosensory feedback; functional balance; gait performance; rehabilitation; four square step test

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control-Vibration (Active Comparator): Participants were assessed before and after 60 days of no additional intervention to any ongoing treatment, after seven days of washout, and after receiving 60 days of vibrotactile ground-contact feedback.
  Interventions: Device: vibrotactile ground-contact feedback
- Vibration-Control (Active Comparator): Participants were assessed before and after receiving 60 days of vibrotactile ground-contact feedback, after seven days of washout, and after 60 days of no additional intervention to any ongoing treatment.
  Interventions: Device: vibrotactile ground-contact feedback

INTERVENTIONS:
Device: vibrotactile ground-contact feedback — Suralis®, Saphenus Medical Technology (Baden, Lower Austria, Austria)

SUMMARY:
Prosthetics research has grown recently, focusing on bionic approaches that restore bodily functions with technical aids. One method involves using prostheses with feedback systems, which measure physical parameters and provide additional information to the user. Saphenus has developed a feedback system called Suralis© that transfers pressure signals from the prosthetic sole to another body region. This clinical investigation aimed to determine if this system improves gait stability and walking. The study analyzed changes in gait and functional balance and gathered patient-reported measures to evaluate the quality of life.

This research was open to individuals who have undergone below-knee amputation but no targeted re-innervation surgery and use prosthetics. Participants received the Suralis© feedback system, and the investigators assessed their walking activities. The system measures prosthetic foot sole pressure and converts it into digital signals, triggering vibration stimuli during the stance phase of walking. The investigators collected gait analyses and patient feedback to assess the impact of the feedback system on prosthetic management. The results will help us understand the benefits and effectiveness of this technology for people with amputation.

DETAILED DESCRIPTION:
The investigators conducted a prospective, unblinded crossover trial to compare the effectiveness of a vibration intervention with no intervention. Participants were randomly assigned to one of two sequences: vibration intervention followed by no intervention or vice versa. The intervention involved using the Suralis© vibrotactile ground-contact feedback system for 60 days. The system transmitted ground contact information to the residual lateral thigh, providing sensory feedback. During the control phase, participants received no additional intervention. The washout period lasted seven days. The study collected data during four visits, assessing gait and patient-reported measures. Bayesian generalized linear mixed models were used for data analysis, considering fixed effects (intervention, sequence, and period) and random effects (individuality).

ELIGIBILITY:
Inclusion Criteria:

* male, female, and diverse individuals
* unilateral transtibial amputation
* at least 18 months post surgery
* walking without aids possible
* signed informed consent form

Exclusion Criteria:

* insufficient thigh sensation to distinguish between the two closest vibrotactile actuators
* an acute event that restricts the walking ability
* interfering lesions or painful conditions
* undergone targeted re-innervation surgery
* poor stump condition
* used a non-modular prosthesis
* used a prosthesis in poor condition
* conditions preventing safe participation or interfering with study objectives
* not able to not comply with the protocol

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-05-06 (Actual)

PRIMARY OUTCOMES:
Affected leg stance time treatment-change difference | Difference between the within-period changes of the 60-day control (C) and vibration (V) periods of the randomized controlled crossover trial, i.e., V(post - pre) - C(post - pre); three tries each assessment day
  Stance time of the prosthetic leg during walking over level ground and on a 518 cm instrumented walkway at a self-selected speed

SECONDARY OUTCOMES:
Gait speed treatment-change difference | Difference between the within-period changes of the 60-day control (C) and vibration (V) periods of the randomized controlled crossover trial, i.e., V(post - pre) - C(post - pre); three tries each assessment day
  Average speed of walking over level ground and on a 518 cm instrumented walkway at a self-selected speed
Unaffected leg step length treatment-change difference | Difference between the within-period changes of the 60-day control (C) and vibration (V) periods of the randomized controlled crossover trial, i.e., V(post - pre) - C(post - pre); three tries each assessment day
  Step length of the non-prosthetic leg during walking over level ground and on a 518 cm instrumented walkway at a self-selected speed
Quality of life score treatment-change difference | Difference between the within-period changes of the 60-day control (C) and vibration (V) periods of the randomized controlled crossover trial, i.e., V(post - pre) - C(post - pre); once each assessment day
  EuroQol (EQ) 5-Dimension (5D) 3-Level (3L) version, visual analog scale (VAS)
Adverse effects frequency treatment difference | Difference in the event frequency during the 60-day control (C) and vibration (V) periods of the randomized controlled crossover trial, i.e., V - C; once each assessment day
  Patient diary documentation and interview regarding adverse effects
Timed up and go test time treatment-change difference | Difference between the within-period changes of the 60-day control (C) and vibration (V) periods of the randomized controlled crossover trial, i.e., V(post - pre) - C(post - pre); three tries each assessment day
  Stand up, walk 3 m, turn around, and sit down
2 min walk test distance treatment-change difference | Difference between the within-period changes of the 60-day control (C) and vibration (V) periods of the randomized controlled crossover trial, i.e., V(post - pre) - C(post - pre); once each assessment day
  Walking distance in meters within a 2 min time frame
Four square step test time treatment-change difference | Difference between the within-period changes of the 60-day control (C) and vibration (V) periods of the randomized controlled crossover trial, i.e., V(post - pre) - C(post - pre); three tries each assessment day
  Do and reverse four steps over 90 cm long canes arranged in a cross configuration on the ground

CONTACTS AND LOCATIONS:
Overall Officials: Gerfried Peternell, MD, Principal Investigator — Ludwig Boltzmann Institute for Traumatology, The Research Center in Cooperation with the AUVA
Locations (1):
- Ordination Dr. Wolfgang Schaden, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that underlie results in the main publication
Supporting Information: Analytic Code
Time Frame: At the time of acceptance in a scientific journal
Access Criteria: The investigators aim to provide broad, equitable, and maximally open access to the dataset and their metadata free of charge in a timely manner after acceptance, consistent with legal and ethical limits required to maintain privacy and confidentiality, tribal sovereignty, and protection of other sensitive data.
URL: https://gitfront.io/r/haripen/6ZQ4pngRwEWa/Safety-Efficacy-vibrotactile-feedback-patients-lower-limb-amputation/

REFERENCES:
- [Derived] Penasso H, Peternell G, Schultheis R, Pitschl A, Leskovar R, Gardetto A, Ernst J, Schmid-Zalaudek K, Schaden W. Safety and efficacy of vibrotactile feedback for adults with transtibial amputation: A randomized controlled cross-over trial. Clin Biomech (Bristol). 2025 Apr;124:106443. doi: 10.1016/j.clinbiomech.2025.106443. Epub 2025 Feb 10. PMID 40054381